CLINICAL TRIAL: NCT06660589
Title: Feasibility Study of Telerehabilitation for People with Chronic Obstructive Pulmonary Disease in Nuuk: Evaluation and Adaptations for Future Rollout Across Greenland
Brief Title: Feasibility Study of Telerehabilitation for People with Chronic Obstructive Pulmonary Disease in Nuuk
Status: Not yet recruiting | Type: Observational
Sponsor: Steno Diabetes Center Greenland (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-20410; NNF20SA0064190 (Other Grant/Funding Number: Novo Nordisk Foundation)
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Greenland; COPD; telerehabilitation; feasibility
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- People with COPD: People with COPD

SUMMARY:
Chronic obstructive pulmonary disease, or COPD, is a major global health issue. It can make people ill, impact their quality of life, and increase their use of healthcare services. In some parts of Greenland, it can be particularly challenging to manage COPD due to the distance to healthcare assistants, nurses, or doctors. Telerehabilitation, which allows people to receive treatment online, could be a good solution.

This project aims to explore how we can best support COPD patients in Nuuk through an online rehabilitation program. The program functions as a pilot study, where we examine how it can be adapted and scaled across Greenland and to patients with other conditions. We will assess how well the program meets patients' needs and determine what adjustments are necessary to improve it.

The study will include 10 individuals with COPD living in Nuuk. They will receive training materials and have an initial meeting with a physiotherapist to set goals. For 10 weeks, they will participate in online training sessions twice a week. Through their feedback, we hope to identify ways to make the program more effective and tailored.

Before the training program begins, participants will have various health metrics measured, complete a questionnaire, and perform a physical test. This will be repeated after the training program is completed to assess any changes in the participants.

We hope that the results will provide insights into improving the treatment of COPD patients and guide necessary adjustments for future rollout across Greenland and to other disease groups. All participants will provide consent for their involvement, and their data will be treated anonymously.

DETAILED DESCRIPTION:
In this study, data will be collected at multiple time points relative to when participants are enrolled:

* Baseline data collection occurs before the intervention begins. Participants will undergo an initial consultation via PUISA, where various assessments (such as the Sit-to-Stand test, CAT score, MRC score, and other health measurements) will be performed. Additionally, participants will fill out a questionnaire and have their physical condition tested.
* Post-intervention data collection occurs after the 10-week training program has concluded. During this final evaluation, the same parameters assessed at baseline (physical condition, CAT questionnaire, etc.) will be measured again. Participants will also provide feedback through qualitative interviews, focusing on their experiences with the program.

Thus, data will be collected both before (pre-intervention) and after (post-intervention) the 10-week telerehabilitation program to evaluate changes and gather feedback.

Sampling method:

The study will employ purposive sampling to select participants who meet specific criteria, such as having a certain level of illness or the ability to participate in a telerehabilitation program. Sampling will be conducted based on age, sex, and degree of illness to ensure a well-defined and relevant participant group.

ELIGIBILITY:
Inclusion Criteria:

* Residing in Nuuk
* Has access to a computer/phone and the internet
* Understands Danish and can participate in a Danish dialogue
* Motivated to participate in online training
* Post-bronchodilator FEV1/FVC ratio below 0.7, and FEV1 below 80% of predicted value
* MRC score of 2 or higher

Exclusion Criteria:

* Unstable angina pectoris
* Hemodynamically significant aortic stenosis
* Physical or psychological condition that prevents benefit from a video consultation, e.g., deafness, muteness, or blindness
* Exacerbation within 6 weeks, lung infection, or other factors that affect the results of a lung function test

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ten individuals diagnosed with COPD and followed at Queen Ingrid's Hospital in Nuuk, Greenland will be identified through electronic medical records.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility criteria: Recruitment | From enrollment to the end of the intervention at 10 weeks.
  How quickly can we recruit participants? What factors hinder patients from participating? Which methods work best to attract patients?
Feasibility criteria: Adherence | From enrollment to the end of the intervention at 10 weeks.
  Active participation will be assessed through attendance rates in the twice-weekly online sessions and adherence to the weekly self-guided session. Motivation and involvement will be gauged by tracking whether participants maintain consistent engagement or drop off over time. Completion of the full 10-week telerehabilitation program will serve as a key indicator of sustained involvement. No-shows and attendance will also be closely monitored.
Feasibility criteria: Acceptability | From enrollment to the end of the intervention at 10 weeks.
  Participants will be asked about their experiences with the video consultation app and other digital tools. They will also provide feedback on the relevance of the telerehabilitation program content in relation to their expectations and needs. Key questions will assess whether participants understood the material and how the technology and content could be improved for better engagement and effectiveness.
Feasibility criteria: Technical challenges | From enrollment to the end of the intervention at 10 weeks.
  Participants will be asked about the quality of their internet connection during sessions, focusing on whether they had reliable access to high-speed internet. They will also assess the functionality of the video consultation app and other digital tools, providing insights into usability and ease of navigation. The study will evaluate any challenges participants faced related to the devices they used for the program. Additionally, participants will provide feedback on the audio and video quality during sessions, noting any issues that may have impacted communication and engagement.

SECONDARY OUTCOMES:
Chair Stand Test (CST) | At enrollment and at the end of the intervention at 10 weeks.
  The CST is designed to assess an individual's ability to perform sit-to-stand movements, which are essential for daily activities such as getting up from a chair, rising from a bed, and maintaining independence.
COPD Assessment Test (CAT) | At enrollment and at the end of the intervention at 10 weeks.
  The CAT is used to evaluate the severity of COPD symptoms and their effect on the patient's health status and quality of life. It helps healthcare professionals monitor disease progression and the effectiveness of treatment interventions.
Smoking status | At enrollment and at the end of the intervention at 10 weeks.
  "Do you currently smoke cigarettes?" (Yes/No) "How many cigarettes do you smoke per day?"
Physical activity | At enrollment and at the end of the intervention at 10 weeks.
  measured by number of daily steps